CLINICAL TRIAL: NCT06532435
Title: A Clinical Study on the Effect of DHA & ARA Candy on the Cognitive Improvement in Preschool Children of 2-6 Years Old
Brief Title: A Clinical Study on the Effect of DHA & ARA Candy on the Cognitive Improvement in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Sibote Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-RD-06-SBT-001
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Change
Keywords: WISC-IV; Cognitive Ability; DHA; ARA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DHA & ARA Candy (Other): Sibot DHA algal oil ARA gelainzed Candy, each containing DHA 100 mg + ARA 100 mg
  Interventions: Dietary Supplement: DHA & ARA Candy

INTERVENTIONS:
Dietary Supplement: DHA & ARA Candy — Parpicipants need to eat 1-2 candy daily, for 4 consective weeks

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness of DHA (docosahexaenoic acid) & ARA (arachidonic acid) Candy on the cognitive development of preschool children (2-6 years old). The main questions it aims to answer are:

- Does DHA & ARA Candy improve the cognitive ability in terms of Wechsler Intelligence Scale for Children 4th edition-Chinese version (WISC-IV-Chinese)?

Researchers will administer the WISC-IV-Chinese following the guidelines strictly and analyze the score to conclude whether the DHA & ARA is effective to improve the cognitive ability of preschool childchildren.

Participants will eat 1-2 candy (each contains 100mg DHA and 100mg ARA) daily for 4 consecutive weeks and take the WISC-IV-Chinese test for three times according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 2-6 years old
* Healthy children of normal development, without gender restrictions, with a male to female ratio of more than 40%;
* During the trial period, participants agree not to take any medications, supplements, or other nutritional products containing DHA and ARA;
* Parents or legal guardians (at least one party) have signed an informed consent form, voluntarily participating in this study and complying with the study design;
* Willing to not participate in other interventional nutritional studies during the trial period;
* Capable of fully understanding the nature, purpose, benefits, and potential risks and side effects of this study.

Exclusion Criteria:

* Allergic to dairy products;
* Severely intolerant to milk dairy products;
* Unable to provide written informed consent;
* During the screening period, or within the past two weeks, has used antibiotics;
* Currently taking therapeutic medications;
* The volunteer has any of the following medical histories or has been nutritionally diagnosed with any of the following diseases: significant gastrointestinal dysfunction, liver, kidney, endocrine, blood, respiratory, or cardiovascular diseases, which may affect the assessment of the trial's effects;
* Suffering from any gastrointestinal dysfunction or gastrointestinal disease. For example, but not limited to: Irritable Bowel Syndrome (IBS), enteritis, ulcerative colitis, celiac disease, irritable bowel syndrome;
* Has a history of hospitalization within the past 3 months;
* According to the researcher's judgment, currently frequently using medications that may affect gastrointestinal function or the immune system.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Change of scale of WISC-IV-Chinese asssessment in 2 weeks | base day 0, week 2
  Change of scale of WISC-IV-Chinese (Wechsler Intelligence Scale for Children 4th edition-Chinese version). The WISC-IV-Chinese is an individually administered and norm-referenced instrument designed to measure intelligence for Chinese children. The WISC-IV contains 10 core subtests and five additional subtests. These are summed into a four-index score and one FSIQ, which ranges from the lowest (40) to the highest (160) points.
Change of scale of WISC-IV-Chinese asssessment in 4 weeks | base day 0, week 4
  Change of scale of WISC-IV-Chinese (Wechsler Intelligence Scale for Children 4th edition-Chinese version). The WISC-IV-Chinese is an individually administered and norm-referenced instrument designed to measure intelligence for Chinese children. The WISC-IV contains 10 core subtests and five additional subtests. These are summed into a four-index score and one FSIQ, which ranges from the lowest (40) to the highest (160) points.

SECONDARY OUTCOMES:
Change of Conners TRS score | base day 0, week 2, week 4
  Change in TRS (Conners' Teacher Rating Scale, TRS ) score over time during the intervention. The Teacher Rating Scales (TRS) are used to measure adaptive and problem behaviors in the preschool or school setting. Teachers or other qualified observers can complete forms at three age levels-preschool (ages 2 to 5), child (ages 6 to 11), and adolescent (ages 12 to 21). The Conners' Teacher Rating Scale we used is a 28-item instrument used to assess children's behavior, each item has four-choice options: 0 = Not True at All (Never, Seldom), 1 = Just a Little True (Occasionally), 2 = Pretty Much True (Often, Quite a Bit), and 3 = Very Much True (Very Often, Very Frequent). The total score ranges from 0 to 54; the smaller the score, the better the behavior.
Number of sick leave days | base day 0, week 2, week 4
  Number of sick leave days of participants during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — Raison Biotech Group
Locations (1):
- Raison Biotech Group Shanghai Lab, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The abstract of the study result will be shared via a public web link
Supporting Information: CSR
Time Frame: The abstract will be available in early November, 2024, and there is no end date for the sharing unless further notice.
Access Criteria: The study result is available to access for the public via the following link http://www.raisonbiotech.com/Data/24-RD-06-SBT-001-Abstract.pdf